CLINICAL TRIAL: NCT00001989
Title: A Randomized Phase II Efficacy, Activity and Safety Study of GLQ223 Alone and in Combination With Zidovudine in Symptomatic HIV-Infected Patients Without Prior Treatment With GLQ223 or Trichosanthin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genelabs Technologies (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 106A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-10

CONDITIONS: HIV Infections
Keywords: Trichosanthin; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Trichosanthin; Zidovudine

INTERVENTIONS:
Drug: Trichosanthin
Drug: Zidovudine

SUMMARY:
This study involves GLQ223 administration to patients who have not previously been exposed to it, but who have received at least 9 months of zidovudine therapy. Efficacy evaluations will include survival, opportunistic infections, T4 cell count, and assessments of viral load.

DETAILED DESCRIPTION:
The study will involve the randomization of patients with 200-500 T4 cells and AIDS or ARC to one of three treatment arms: zidovudine alone, GLQ223 alone, or GLQ223 plus zidovudine. Patients randomized to receive GLQ223 will receive an infusion every three weeks for 45 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine, trimethoprim/sulfamethoxazole, or dapsone for PCP prophylaxis.
* Chronic suppressive therapy for the following infections:

Toxoplasmosis (pyrimethamine, sulfadiazine, or clindamycin). Cryptococcosis (fluconazole). Candidiasis (ketoconazole). Herpes simplex virus (acyclovir). Mycobacterium avium (isoniazid, clofazimine, amikacin, rifampin, rifabutin, ethambutol, or other drug with written permission of the sponsor).

Required:

* Patients whose CD4+ count falls below 200 at two consecutive measurements must receive prophylaxis for PCP and any other clinically indicated conditions.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* An active AIDS-defining opportunistic infection.
* Evidence of AIDS dementia complex or active neurologic disease, including progressive multi-focal leukoencephalopathy (PML), poorly controlled seizure disorder or active CNS infection.
* Any condition which in the Investigator's opinion is sufficient to prevent adequate compliance with the study.

Concurrent Medication:

Excluded:

* Therapeutic agents specific for HIV disease that have not received FDA approval.
* Biologic response modifiers, including interferon, interleukin-2 (IL-2), and leukocyte stimulating hormones (GM-CSF, G-CSF).

Patients with the following are excluded:

* An active AIDS-defining opportunistic infection.
* Evidence of AIDS dementia complex or active neurologic disease, including progressive multi-focal leukoencephalopathy (PML), poorly controlled seizure disorder or active CNS infection.
* Participation in other clinical studies, including investigational therapy of HIV infection.
* Any condition which in the Investigator's opinion is sufficient to prevent adequate compliance with the study.
* History of prior use of GLQ223 or trichosanthin or presence of anti-GLQ223 serum IgG antibody as measured by Western blot.
* Inability to provide written informed consent.

Prior Medication:

Excluded:

* History of prior use of GLQ223 or trichosanthin or presence of anti-GLQ serum IgG antibody as measured by Western blot.

Excluded within 30 days prior to enrollment:

* Use of unapproved therapeutic agents specific for HIV disease, including ddC.
* Use of biologic response modifiers, including interferon, interleukin-2, and leukocyte stimulating hormones (GM-CSF, G-CSF).

Patients have the following:

* HIV positive by ELISA with confirmation by Western blot.
* Symptomatic with AIDS-Related Complex or AIDS by CDC classification.
* History of zidovudine therapy at a dose equal to or more than 300 mg daily for at least 9 consecutive months immediately prior to entry into study.
* CD4 count equal to or more than 200 and equal to or less than 500 (mean of 2 readings one week apart).
* Ability to give informed consent.

Required:

* Zidovudine therapy at a dose equal to or more than 300 mg daily for at least 9 months immediately prior to entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - ViRx Inc, San Francisco, California
  - Dr Larry A Waites, San Francisco, California
  - Saint Francis Mem Hosp, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Northwestern Univ, Chicago, Illinois
  - Saint Vincent's Hosp and Med Ctr, New York, New York

REFERENCES:
- [Background] Byers VS, Levin AS, Malvino A, Waites L, Robins RA, Baldwin RW. A phase II study of effect of addition of trichosanthin to zidovudine in patients with HIV disease and failing antiretroviral agents. AIDS Res Hum Retroviruses. 1994 Apr;10(4):413-20. doi: 10.1089/aid.1994.10.413. PMID 7915124
- [Background] Waites AL, Klimas N, Yangco B, Chew T, Lang W, Von Roenn J, Torres G, Gorelick KJ, Kahn JO. Final report of a randomized phase II study of GLQ223 in AIDS and ARC. Program Abstr Intersci Conf Antimicrob Agents Chemother. 1994 Oct 4-7:61